CLINICAL TRIAL: NCT03071458
Title: Translating Molecular Classifications and Genetic Alterations of Hepatocellular Carcinoma in Clinical Care (MUTHEC Project)
Brief Title: Mutational Landscape in Hepatocellular Carcinoma
Acronym: MUTHEC
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C 16-71
Record Dates: First submitted 2017-01-02; First posted 2017-03-07 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2017-03

CONDITIONS: HepatoCellular Carcinoma; Cirrhosis
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 224 tumor (HCC) and 224 non tumor samples from liver transplantation 129 tumor (HCC) and 129 non tumor samples from radio frequency ablation 342 tumor (HCC) and 342 non tumor samples from liver resection 40 tumor (HCC) and 35 non tumor samples from biopsies of advanced HCC 277 plasmas of 78 patients for circulating tumor DNA analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with HCC: The cohort is composed of patients with HCC with available tumor and non tumor samples collected retrospectively. These patients have HCC of different stages (localized and advanced stages) It is an observational retrospective study.

SUMMARY:
The MUTHEC project aims to describe the mutational and transcriptomic landscape of HCC treated by curative treatments (resection, radio frequency ablation, transplantation) as well as advanced HCC together with the analysis of circulating tumor DNA.

DETAILED DESCRIPTION:
Scientific context

Hepatocellular carcinoma (HCC) is one of the leading causes of cancer death worldwide. A transcriptomic classification (G1-G6) described by our lab have underlined the heterogeneity of HCC and identified relationship between transcriptomic group and clinical and genetic features. Recently, a diagnostic and molecular algorithm has been developed to perform the diagnosis of benign and malignant hepatocellular tumors and assess the prognosis of resected HCC. Whole-exome sequencing has also identified new oncogenes and tumor suppressor genes in HCC. However, these studies have focused on HCC treated by liver resection and they have to be validated in biopsy and surgical pieces in larges series of patients treated by resection, liver transplantation and radiofrequency ablation (RFA). In addition, next-generation sequencing allows to sequence circulating tumor DNA in plasma of patients with advanced cancer but it has never tested in patients with HCC.

Description of the project The MUTHEC project involves 4 teams in France and aims to perform translation of molecular and genetic classification of HCC in clinical care.

First, the investigators want to draw a genetic landscape of HCC in different clinical settings. The investigators will sequence 30 genes, previously identified by whole exome sequencing, in a series of 120 HCC treated by RFA, 200 HCC treated by liver transplantation and 40 advanced HCC. The investigators also aim to validate our diagnostic and prognostic molecular algorithm (56 genes including the prognostic 5-gene score using quantitative RT-PCR) in different clinical settings and test their uses in formalin-fixed, paraffin-embedded (FFPE) tissues. In addition, the investigators will test surrogate markers of genetic alterations and oncogenic pathways using immunohistochemistry in these series of tumors. All the HCC will be reviewed by expert pathologist in order to perform genotype/phenotype classification. Lastly, the investigators want to conduct a pilot study to sequence circulating tumor DNA. The investigators will use next generation sequencing to detect in the plasma the somatic mutation observed in tumor biopsy. It will allow a non-invasive diagnosis of tumor mutation in the plasma of patients before and after treatment by RFA.

Expected results The investigators aim to extend our knowledge of HCC genetic alterations in the different types of curative treatment (resection, liver transplantation and RFA) and in advanced HCC. In addition, the investigators want to translate this classification using immunohistochemistry to facilitate it uses in routine. These results will be used in the future to identify subgroups predict to response to targeted treatment. In addition, the investigators will validate our diagnostic and prognostic molecular signature in different clinical situation and in FFPE samples. Assessment of prognosis after curative treatment will help to stratify adjuvant treatment in the future and guide therapeutic decision. Finally, sequencing circulating tumor DNA would allow monitoring somatic mutations ("liquid biopsy") after curative treatment and under the selective pressure of targeted therapies.

ELIGIBILITY:
Inclusion Criteria:

* Written consent of the patient according to the French Law: the French Liver Biobanks network - AFAQ NF S96-900 and Hepatobio bank
* Histologically proven hepatocellular carcinoma
* Available frozen samples
* HCC assessible to a curative treatment (Treated by resection, liver transplantation, radio frequency ablation) or advanced HCC with available biopsy

Exclusion Criteria:

* Less than 18 years old
* Pregnancy at the date of the sample
* Parafinn embedded tissue only available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with hepatocellular carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 808 (Actual)
Dates: Start 2008-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Genetic and transcriptomic landscape | Up to 3 years
  Identification of the main genetic driver and transcriptomic subgroups among a large panel of HCC

SECONDARY OUTCOMES:
Translation in immunohistochemical markers | Up to 3 years
  The investigators aim to translate the major genetic drivers and oncogenic pathway dysregulated in HCC using immunohistochemistry. The investigators will test surrogate markers of the main genetic alterations and activation of oncogenic pathway using immunohistochemistry in HCC extensively reviewed by expert pathologists.
Detection and sequencing of circulating tumor DNA as a liquid biopsy in HCC | Up to 3 years
  The aim is to conduct a pilot and innovative study to detect mutations in DNA circulating in peripheral blood (ctDNA) in patients with early and advanced HCC. The results will be compared to that obtained in the tumor.
Validation of the molecular classification by integrative analysis | Up to 3 years
  At the end, the investigators aim to perform an integrative analysis of all the data generated by tumor analyses and collected in a database using the various approaches: clinical data, pathological and immunohistochemical features, molecular classification and genetic alterations.

CONTACTS AND LOCATIONS:
Overall Officials: jessica zucman-rossi, Md,Phd, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France; jean-charles Nault, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- INSERM, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Blaise L, Ziol M, Campani C, Ganne-Carrie N, Nahon P, Nkontchou G, Zucman-Rossi J, Del Pozo L, Barget N, Boros C, Desjonqueres E, Demory A, Grando V, Pescatori L, Seror O, Sutter O, Nault JC. Utility of tumor and non-tumor biopsies during percutaneous radiofrequency ablation for hepatocellular carcinoma. JHEP Rep. 2025 Apr 22;7(9):101430. doi: 10.1016/j.jhepr.2025.101430. eCollection 2025 Sep. PMID 40823168